CLINICAL TRIAL: NCT03603691
Title: A Single-centre, Prospective, Cross-sectional Study to Evaluate the Reliability and Validity of the Modified Manual Muscle Test for Persons With Multiple Sclerosis) (MS)
Brief Title: Study to Evaluate the Reliability and Validity of the Modified Manual Muscle Test for Persons With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanco van der Maas (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); Physiotherapie Langmatten Binningen, Switzerland (Unknown); Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Nanco van der Maas, Principle Investigator, Institut fuer Physiotherapieforschung
Organization: Institut fuer Physiotherapieforschung (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2018-01103; me16Kappos3
Record Dates: First submitted 2018-06-19; First posted 2018-07-27 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Prospective, cross-sectional and test-retest
Who Masked: Outcomes Assessor
Masking Description: the outcome assessors will be blinded for the results of other assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Modified Manual Muscle Test (Active Comparator): The MMMT will be tested in a test-retest design
  Interventions: Diagnostic Test: Modified Manual Muscle Test; Diagnostic Test: BMRC manual muscle test; Diagnostic Test: MicroFET2 handhold dynamometer; Diagnostic Test: Modified Tardieu Scale; Diagnostic Test: Fatigue Scale for Motor and Cognitive Functions; Diagnostic Test: numeric rating scale Fatigue
- Neurostatus BMRC (Active Comparator): The Neurostatus BMRC measures Strength and will be used in a test-retest design
  Interventions: Diagnostic Test: Modified Manual Muscle Test; Diagnostic Test: BMRC manual muscle test; Diagnostic Test: MicroFET2 handhold dynamometer; Diagnostic Test: Modified Tardieu Scale; Diagnostic Test: Fatigue Scale for Motor and Cognitive Functions; Diagnostic Test: numeric rating scale Fatigue
- MicroFET2 (Active Comparator): The MicroFET2 is a hand held dynamometer to measure strength
  Interventions: Diagnostic Test: Modified Manual Muscle Test; Diagnostic Test: BMRC manual muscle test; Diagnostic Test: MicroFET2 handhold dynamometer; Diagnostic Test: Modified Tardieu Scale; Diagnostic Test: Fatigue Scale for Motor and Cognitive Functions; Diagnostic Test: numeric rating scale Fatigue

INTERVENTIONS:
Diagnostic Test: Modified Manual Muscle Test — Manual Muscle Testing Grading System from 0=No visible or palpable contraction to 5= full range of movement against gravity, maximal resistance
Diagnostic Test: BMRC manual muscle test — muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle
Diagnostic Test: MicroFET2 handhold dynamometer — MicroFET 2 Handheld Dynamometer is a force evaluation testing device to evaluate the strength of various muscle groups
Diagnostic Test: Modified Tardieu Scale — Modified Tardieu Scale is to measure if there is spasticity present in a person's muscle and its response to movement
Diagnostic Test: Fatigue Scale for Motor and Cognitive Functions — Measures cognitive and motor fatigue for people with MS
Diagnostic Test: numeric rating scale Fatigue — visual analog scale that uses a scalar numbering system to objectify a patient's fatigue (0 = no fatigue; 10 = most extreme fatigue)

SUMMARY:
Many patients with multiple sclerosis (MS) are treated with physiotherapy. Muscle weakness is a common symptom. It can be evaluated with a variety of muscle function tests. In MS patients, testing muscle function can be confounded by many factors, such as spasticity and ataxia, which are not considered by the existing tests and may cause biased test results. Steinlin Egli described a Modified Manual Muscle Test (MMMT) that considers spasticity and may provide a more reliable and valid muscle function test for MS patients.

The investigators aim to evaluate the inter- and intra-rater reliability of the Modified Manual Muscle Test in MS and evaluate the validity of the Modified MMT according to the criteria of the 6 level British Medical Research Council (BMRC) manual muscle test and the microFET2 handhold dynamometer.

DETAILED DESCRIPTION:
Background In Switzerland, many patients with multiple sclerosis (MS) are treated with physiotherapy. Muscle weakness is a common symptom. Particularly in progressive disease courses, motor dysfunction is a major contributor to the reduced mobility and quality of life. Therefore, improving the motor dysfunction is an important goal for therapy and is evaluated with a variety of muscle function tests. The 6 level British Medical Research Council (BMRC) manual muscle test is the most widely used test in MS and is a part of the Neurostatus-Expanded Disability Status Scale (EDSS) assessment, which has been adopted as the standard in most of the pivotal trials that have led to the approval of the current MS treatments. In MS patients, testing muscle function can be confounded by many factors, such as spasticity and ataxia, which are not considered by the existing tests and may cause biased test results. Steinlin Egli described a Modified Manual Muscle Test (MMMT) that considers spasticity and may provide a more reliable and valid muscle function test for MS patients.

Aim of the study is to evaluate the inter- and intra-rater reliability of the Modified Manual Muscle Test in MS and evaluate the validity of the Modified MMT according to the criteria of the Neurostatus BMRC manual muscle test and the microFET2 handhold dynamometer.

Methods This is a single-centre, prospective cross-sectional study with a test-retest design. The Neurostatus BMRC manual muscle test and the microFET2 hand held dynamometer are used as the criteria. The primary endpoint is the ordinal MMMT level. The intra-class correlation coefficient (ICC) of the ranked MMMT levels will be estimated. The investigator aims to show that the MMMT results are clinically relevant with a high level of ICC.

The secondary endpoints include the Neurostatus BMRC levels, the muscle strength as measured by the microFET2 dynamometer and fatigue using a numeric rating scale (NRS). Subgroup analyses will determine whether the MMMT is less sensitive to the influence of spasticity than the Neurostatus BMRC.

28 patients with MS will be tested in 2 days. In each day, six examiners will test seven patients in the morning and seven patients in the afternoon. Three MS-therapists from the Specialized Group Physiotherapy in MS and three neurologists from the Department of Neurology at the University Hospital Basel will be tester. All examiners will be blinded to the results of the other examiners. All test persons will be blinded to their test results. First, the patient will rate his fatigue using the NRS. Muscle function will be tested with the microFET2 and spasticity will be assessed using the modified Tardieu Scale. Then, the first round of manual testing will be executed. After each test, there will be a break that is long enough for the patients to recuperate. The order of the examiners will be randomized. The retest round will proceed in a different order. Finally, spasticity will be tested again using the modified Tardieu Scale, and the patients will rate their fatigue.

Statistical Analysis The study data will be analysed using the internet-based program R. The descriptive statistics will describe the sample characteristics. The inter-rater reliability will be estimated by the ICC of the MMMT ranks. The ICC will be estimated by a two-way random-effects ANOVA and reported with 95% CI. If the lower limit of the CI is larger than the pre-specified clinically relevant ICC margin, the MMMT will be considered a reliable tool for evaluating muscle strength in MS patients.

The inter-rater reliability the Neurostatus BMRC will be estimated similarly by the ICC. The ICC of both tests will be compared. The test-retest reliability of the MMMT and Neurostatus BMRC will be estimated using two-way random-effects ANOVA and will be reported by ICC estimates. The influence of potential fatigue will be analysed by plotting the test and retest results against the NRS and investigating the associations and interactions using a linear mixed effects model. The pairwise correlations of the MMMT and the Neurostatus BMRC with the microFET2 will be graphically analysed (scatterplots and/or boxplots), and Spearman's ρ will be calculated. The primary and secondary analyses will be repeated for subgroups with high and low spasticity patients to compare the sensitivity of the MMMT and Neurostatus BMRC to spasticity.

Expected results: The investigators expect the MMMT for MS to be a reliable and valid manual muscle function test that can be used in the evaluation of the long-term treatment of MS patients with physical therapy.

ELIGIBILITY:
Inclusion Criteria

* diagnosed with MS according to the McDonald criteria
* EDSS between 0 and 6.5
* older than 18 years of age.

Exclusion Criteria:

* An acute episode of MS within 3 months prior to the testing,
* grave cognitive changes
* distinct fatigue
* a history of current back, neck or elbow pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Inter-rater reliability Modified Manual Muscle Test | Baseline
  The primary endpoint is the MMMT level. The ordinal levels (2+, 3-, 3, 4-, 4, 4+ and 5) will be transformed to ranks (1-7), and the intra-class correlation coefficient (ICC) of the ranked MMMT levels will be estimated. The aim is to show that the MMMT results are at a clinically relevant - thus high - level of ICC (that is a pre-specified, clinically relevant level the ICC margin).
  The null hypothesis is that the lower limit of the 95% confidence interval (CI) of the ICC is smaller than or equal to the ICC margin. The alternative hypothesis is that the lower limit of the 95% CI of the ICC is larger than the ICC margin.
  If the lower limit of the CI is larger than the ICC margin, the MMMT will be considered a reliable tool for evaluating muscle strength in MS patients.

SECONDARY OUTCOMES:
Intra-rater reliability Modified Manual Muscle Test | Baseline- Baseline plus 4 hours
  The intra-rater reliability will be evaluated by comparing the test results of two tests (test-retest), which will be executed by the same tester. The two tests will be executed on the same day within 4 hours. The intra-class correlation coefficient of the ranked MMMT levels (analogue to the primary endpoint) will be used to describe the intra-rater reliability of the MMMT.
Validity of the Modified Manual Muscle Test | Baseline- Baseline plus 4 hours
  The inter-rater reliability of the BMRC will be measured by the ICC. The ICC of the BMRC will be estimated and analysed as previously described for the primary analysis. The ICCs of the MMMT and the BMRC will be compared descriptively.
  The test-retest reliability of the MMMT and the BMRC will be estimated for each rater separately using a two-way random-effects ANOVA, including the patient and "test type" (test/retest) as random effects. The ICC estimates will be reported with the 95% CI and compared descriptively between the raters using the same test and between the tests (MMMT vs BMRC).
  The pairwise correlations of the MMMT and the BMRC with the muscle strength as assessed by the microFET2 will be investigated graphically (scatterplots and/or boxplots). Furthermore, Spearman's rank correlation coefficient will be presented with the corresponding 95% CI and p-values.
Modified Tardieu Scale level | Baseline- Baseline plus 4 hours
  The BMRC has 6 levels, which makes the scale robust and reliable but insensitive to change. In addition, the BMRC does not consider spasticity. The MMMT has 12 levels, which makes it more sensitive, but it also might mean that the scale is less reliable. Because the MMMT considers spasticity, we expect that this compensates for the possible loss of reliability. It is assumed that the MMMT is less sensitive to spasticity than the BMRC. Thus, for patients with a different level of spasticity measured by the Modified Tardieu Scale, both the inter-rater and the test-retest reliability of the MMMT are expected to be equal to those of the BMRC.
  The primary and secondary analyses will thus be repeated for the subgroups of high-spasticity and low-spasticity patients separately (assuming that a reasonable number of patients per subgroup and endpoint are available).

OTHER OUTCOMES:
Bias testing Fatigue | Baseline- Baseline plus 4 hours
  The study may be biased by the multiple testing that cause motor fatigue. The test and retest ratings will be plotted against the respective Numeric Rating Scale fatigue (at the beginning or end of the assessment, respectively) and tested for an overall association and interaction using a linear mixed effects model.

CONTACTS AND LOCATIONS:
Overall Officials: Nico van der Maas, Principal Investigator — Institute for Physiotherapy Research, Biel, Switzerland; Marcus Dsouza, Dr. med., Principal Investigator — University Hospital Basle, Basle, Switzerland; Regula Steinlin Egli, Principal Investigator — Specialized Group Physiotherapy in MS, Binningen, Switzerland
Locations (1):
- Felix Platter Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided